CLINICAL TRIAL: NCT06336473
Title: Evaluation of the Effects of Cross Linking on the Biomechanical Characteristics of Skin Samples From Patients With Classic or Hypermobile Ehlers-Danlos Syndrome
Acronym: SEDSKIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A02097-38
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Intervention Model Description: Single-center study performed on biopsied skin samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin biopsy (Experimental)
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — Samples will be taken under local anaesthetic (after injection of 1 cc of Xylocaine without adrenaline) using a 4 mm diameter dermal biopsy punch. The biopsy will be performed on the buttocks. Fragments are stored in 15-mL polypropylene tubes in PBS at 4°C.

SUMMARY:
The main aim of this study is to evaluate the effect of cross linking on the elasticity of skin samples from patients with non-vascular Ehlers-Danlos Syndrome (hEDS or cEDS).

DETAILED DESCRIPTION:
This is a single-center study based on skin biopsies. The skin biopsies will be taken at the non-vascular Ehlers-Danlos syndromes reference center at the Raymond Poincaré Hospital (Garches), by Dr. Karelle Benistan. This center regularly performs this type of biopsy as part of its routine care, and has set up a fibroblast bank for Genethon (Authorization for biological collection at Genethon: SED BACG n° DC-2021-4628).

Samples will be transported to the Centre de Recherche Saint-Antoine (UMR-S 938) where they will be processed, cut and placed on histological slides.

Atomic force microscopy analyses will be carried out at the Laboratoire de Réactivité de Surface (CNRS/Sorbonne University).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over, having read and signed the consent form for participation in the study
* Patient with classic or hypermobile Ehlers-Danlos syndrome
* Regularly followed-up at the non-vascular Ehlers-Danlos Syndrome Reference Center at Garches Hospital.

Exclusion Criteria:

* Patient under court protection, guardianship or curatorship
* Pregnant or breast-feeding patient
* Patient not affiliated to the French social security system
* Impossibility of giving the subject informed information and/or written informed consent: dementia, psychosis, disturbed consciousness, non-French-speaking patient
* Contraindication to anaesthesia or allergy to local anaesthetic product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-03 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Young's modulus quantification | Day 0
  Atomic force microscopy (AFM), in contact mode, enables force curves to be obtained. The tip no longer scans the surface of the sample, but probes the surface at several indentation points.
  A microlever deflection curve is generated for each indentation point.
  Calculation of Young's modulus is based on Bilodeau's model, in which the tip is assimilated to a pyramid in contact with a flat surface.
  F is the measured force, E the modulus of elasticity, α the face angle of the pyramid, δ the indentation depth and ν the Poisson's ratio of the sample, set at 0.5 (corresponding to an incompressible material).
  Young's modulus will be quantified by AFM

SECONDARY OUTCOMES:
Collagen fibril diameter measurement | Day 0
  Three 2 μm x 2 μm images with at least 100 scan lines will be acquired on each sample and used to describe the intrinsic characteristics of collagen fibrils.
Collagen fibril D-period length measurement | Day 0
  Three 2 μm x 2 μm images with at least 100 scan lines will be acquired on each sample and used to describe the intrinsic characteristics of collagen fibrils.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Maussins-Nollet, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided